CLINICAL TRIAL: NCT02370043
Title: Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Food Effect of KQ-791 in Healthy Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Food-Effect of KQ-791
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kaneq Bioscience Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: KQ-791-01
Record Dates: First submitted 2015-02-18; First posted 2015-02-24 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers; Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Postprandial Period

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- KQ-791 (Experimental): Escalating doses of KQ-791, starting at 15 milligrams
  Interventions: Drug: KQ-791
- KQ-791 (after meal) (Experimental): Single dose of KQ-791 in capsule form, after a meal
  Interventions: Drug: KQ-791 (after meal)
- Placebo (Placebo Comparator): Single dose of placebo matching KQ-791 dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KQ-791 — Capsules administered orally while fasting, in up to 3 periods
  Arms: KQ-791
Drug: KQ-791 (after meal) — Single dose of KQ-791 in capsules, after a meal, in 1 period
  Arms: KQ-791 (after meal)
Drug: Placebo — Capsules, administered orally, in 1 period
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and the effect of food on KQ-791. Each participant may receive up to 3 single doses of KQ-791 (at up to 3 different dose levels) and 1 placebo dose over the course of the study. Up to 6 escalating dose levels may be studied, in two distinct groups or cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-childbearing potential female, which includes post-menopausal female (absence of menses for 12 months prior to drug administration, bilateral oophorectomy or hysterectomy with bilateral oophorectomy at least 6 months prior to drug administration) or surgically sterile female (hysterectomy or tubal ligation at least 6 months prior to drug administration)
* Body Mass Index (BMI) greater than or equal to (≥) 27.0 and less than or equal to (≤) 35.0 kilogram per square meter (kg/m2)
* Healthy as defined by:

  1. absence of clinically significant illness and surgery within last 4 weeks. Participants vomiting within 24 hours pre-dose will be evaluated for upcoming illness/disease
  2. the absence of clinically significant history of neurological, endocrine, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, or metabolic disease
* Male participants who are not vasectomized for at least 6 months, and who are sexually active with non-sterile female partner (sterile female partners include post-menopausal females and surgically sterile females) must be willing to use one of the following acceptable contraceptive methods throughout the study and for 90 days after the last study drug administration:

  1. simultaneous use of a condom, and for the female partner hormonal contraceptives (used since at least 4 weeks) or intra-uterine contraceptive device (placed since at least 4 weeks)
  2. simultaneous use of a male condom, and for his female partner, a diaphragm with intravaginally applied spermicide
* Some degree of insulin resistance, as shown by:

  1. fasting blood glucose ≥95.4 and ≤126 milligrams per deciliter (mg/dL) (equivalent to 5.3 to 7.0 millimoles per liter (mmol/L), respectively) and
  2. fasting triglycerides ≤ 4.0 mmol/L, and/or
  3. Low-Density Lipoprotein Cholesterol (LDL-C) ≤ 6.0 mmol/L
* Capable of consent
* Non-smoker (no use of tobacco products within the last 3 months)

Exclusion Criteria:

* Any clinically significant abnormality or abnormal laboratory test results (other than glucose,triglycerides and LDL-C levels described in inclusion criterion)
* Positive test for hepatitis B, hepatitis C, or Human Immunodeficiency Virus (HIV)
* Evidence of clinically significant hepatic or renal impairment, including Alanine Aminotransferase (ALT) above 1.5x Upper Limit of Normal (ULN), Aspartate Aminotransferase (AST) above 2x ULN, total bilirubin above 2x ULN (total bilirubin accepted up to 2x ULN if direct bilirubin is within normal limits), or Estimated Glomerular Filtration Rate (eGFR) less than (<) 90 milliliters per minute (mL/minute)
* Positive urine drug screen
* History of significant allergic reactions (e.g. angioedema) to any drug.
* Use of any drugs known to induce or inhibit hepatic drug metabolism within the last 30 days
* Positive pregnancy test
* Any reason which, in the opinion of the qualified investigator (QI) would prevent the subject from participating in the study
* Clinically significant electrocardiogram (ECG) abnormalities at screening, or clinically significant personal or family history (in a first-degree relative) of heart diseases, including:

  1. Confirmed corrected QT (QTcF) interval greater than (>) 450 milliseconds (msec) for men and women
  2. Bundle branch blocks and other conduction abnormalities other than mild first degree atrio-ventricular block
  3. Irregular rhythms other than sinus arrhythmia or occasional, rare supraventricular ectopic beats
* History of unexplained syncope
* Family history of unexplained sudden death or sudden death due to long QT syndrome
* T-wave configurations are not of sufficient quality for assessing QT interval
* Clinically significant vital sign abnormalities (systolic blood pressure lower than 90 or over 150 mmHg, diastolic blood pressure lower than 50 or over 95 mmHg, or heart rate less than 50 or over 100 beats per minute (bpm))
* History of significant alcohol abuse within one year prior to screening or regular use of alcohol within six months prior to the screening (regular use of more than three units of alcohol per day for males and more than two units of alcohol per day for females [1 unit = 150 (milliliter) mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]) or positive alcohol breath test
* History of significant drug abuse within the last year or use of soft drugs (such as marijuana) within 3 months prior, or hard drugs (such as cocaine, phencyclidine (PCP) and crack) within the last year
* Participation in a clinical trial involving the administration of an investigational or marketed drug within the last 30 days (90 days for biologics) or concomitant participation in an investigational study
* Use of medication other than topical products without significant systemic absorption:

  1. prescription medication within last 14 days
  2. over-the-counter products within the last 7 days, with the exception of the occasional use of acetaminophen (up to 2 grams (g) daily)
  3. natural health products (e.g. food supplements or herbal supplements) within last 14 days
  4. a depot injection or an implant of any drug within last 3 months
* Donation of plasma within the last 7 days. Donation or loss of blood of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days
* Hemoglobin <128 grams per liter (g/L) (males) and <115 g/L (females) and hematocrit <0.37 L/L (males) and <0.32 L/L (females)
* Breast-feeding participant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email: daniel.bouthillier@Kaneq.ca, Study Director — Kaneq Bioscience
Locations (2):
- Canada (2):
  - Inventiv, Montreal, Quebec
  - inVentiv, Québec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sequence 60 mg/600 mg/Placebo subject discontinued after completion of 600 mg. Sequence Placebo/600 mg/1800 mg subject discontinued after completion of placebo.
Period: Overall Study
Arm/Group | Sequence: 15 mg/Placebo/1200 mg/Placebo (Fed) | Sequence: 15 mg KQ791/195 mg/Placebo/195 mg (Fed) | Sequence: Placebo/195 mg/1200 mg/195 mg (Fed) | Sequence: 60 mg/Placebo/1800 mg | Sequence: 60 mg/600 mg/Placebo | Sequence: Placebo/600 mg/1800 mg
Started | 3 | 3 | 3 | 3 | 3 | 4
Completed | 3 | 3 | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Events (SAEs) Considered by the Investigator to be Related to Study Drug
Time Frame: Baseline to study completion (up to 11 weeks)
Measure: Number; unit: participants
Arm/Group | 15 mg KQ-791 (Fasting) | 60 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fed) | 600 mg KQ-791 (Fasting) | 1200 mg KQ-791 (Fasting) | 1800 mg Kq-791 (Fasting) | Placebo (Fed) | Placebo (Fasting)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 17
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Non-Zero Concentration (AUC0-t)
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8,10, 24, 48, 96, and 144 hours post-dose, and on Day 10 for all dose levels, and on Day 28 for dose level 195 mg; on Days 14 and 28 for dose level 600 mg; and on Days 14, 28, and 56 for dose level 1800 mg
Population: All randomized participants who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute AUC0-t.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 15 mg KQ-791 (Fasting) | 60 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fed) | 600 mg KQ-791 (Fasting) | 1200 mg KQ-791 (Fasting) | 1800 mg Kq-791 (Fasting)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*ng/mL | 34699.23 (44.87) | 95223.95 (32.54) | 358380.52 (36.34) | 110566.98 (17.39) | 721393.21 (32.49) | 1207610.37 (29.83) | 2137673.75 (34.74)

3. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to 24-hour Post-Dose (AUC0-24)
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8,10, and 24 hours post-dose
Population: All randomized participants who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute AUC0-24.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 15 mg KQ-791 (Fasting) | 60 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fed) | 600 mg KQ-791 (Fasting) | 1200 mg KQ-791 (Fasting) | 1800 mg Kq-791 (Fasting)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*ng/mL | 3410.02 (55.50) | 12251.48 (25.11) | 33151.96 (34.63) | 16718.65 (17.76) | 60448.26 (46.92) | 113891.92 (24.54) | 178100.82 (44.64)

4. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC0-inf)
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8,10, 24, 48, 96, and 144 hours post-dose, and on Day 10 for all dose levels, and on Day 28 for dose level 195 mg; on Days 14 and 28 for dose level 600 mg; and on Days 14, 28, and 56 for dose level 1800 mg'
Population: All randomized participants who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute AUC0-inf.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 15 mg KQ-791 (Fasting) | 60 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fed) | 600 mg KQ-791 (Fasting) | 1200 mg KQ-791 (Fasting) | 1800 mg Kq-791 (Fasting)
Number analyzed (Participants) | 5 | 3 | 6 | 2 | 6 | 6 | 6
h*ng/mL | 40581.44 (51.90) | 128600.49 (37.47) | 387934.16 (31.98) | 120230.35 (9.81) | 776014.78 (37.64) | 1311488.40 (29.23) | 2176168.42 (34.65)

5. Secondary Outcome: Maximum Observed Drug Concentration (Cmax)
Time Frame: as for outcome 2
Population: All randomized participants who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 15 mg KQ-791 (Fasting) | 60 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fed) | 600 mg KQ-791 (Fasting) | 1200 mg KQ-791 (Fasting) | 1800 mg Kq-791 (Fasting)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 188.65 (65.96) | 637.51 (29.32) | 1857.08 (45.29) | 923.51 (20.32) | 3238.86 (52.73) | 5828.97 (32.07) | 9418.01 (44.09)

6. Secondary Outcome: Residual Area
Description: calculated as 100*(1- AUC0-t / AUC0-inf)
Time Frame: as for outcome 2
Population: All randomized participants who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute Residual Area.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage residual area under the AUC
Arm/Group | 15 mg KQ-791 (Fasting) | 60 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fed) | 600 mg KQ-791 (Fasting) | 1200 mg KQ-791 (Fasting) | 1800 mg Kq-791 (Fasting)
Number analyzed (Participants) | 5 | 3 | 6 | 2 | 6 | 6 | 6
Percentage residual area under the AUC | 4.59 (107.28) | 11.51 (45.28) | 3.58 (113.37) | 13.23 (50.26) | 4.25 (88.29) | 4.53 (84.07) | 1.55 (47.64)

7. Secondary Outcome: Time to Observed Cmax (Tmax)
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8,10, 24, 48, 96, and 144 hours post-dose, and on Day 10 for all dose levels
Population: All randomized participants who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute Tmax.
Measure: Median (Full Range); unit: Hours
Arm/Group | 15 mg KQ-791 (Fasting) | 60 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fed) | 600 mg KQ-791 (Fasting) | 1200 mg KQ-791 (Fasting) | 1800 mg Kq-791 (Fasting)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours | 4 [2 to 7.99] | 5 [4 to 8] | 4 [3.99 to 48] | 8 [6 to 10] | 5.01 [4 to 8] | 8 [4 to 10] | 7.06 [4 to 8]

8. Secondary Outcome: Elimination Half-Life (T1/2 el)
Time Frame: as for outcome 2
Population: All randomized participants who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute T1/2 el.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | 15 mg KQ-791 (Fasting) | 60 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fed) | 600 mg KQ-791 (Fasting) | 1200 mg KQ-791 (Fasting) | 1800 mg Kq-791 (Fasting)
Number analyzed (Participants) | 5 | 3 | 6 | 2 | 6 | 6 | 6
Hours | 200.67 (16.89) | 196.45 (17.67) | 214.42 (28.77) | 76.86 (22.80) | 219.71 (7.83) | 197.77 (24.28) | 215.58 (12.61)

9. Secondary Outcome: Elimination Rate Constant (Kel)
Time Frame: as for outcome 2
Population: All randomized participants who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute Kel.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour
Arm/Group | 15 mg KQ-791 (Fasting) | 60 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fed) | 600 mg KQ-791 (Fasting) | 1200 mg KQ-791 (Fasting) | 1800 mg Kq-791 (Fasting)
Number analyzed (Participants) | 5 | 3 | 6 | 2 | 6 | 6 | 6
Per hour | 0.0035 (18.9823) | 0.0035 (16.0482) | 0.0032 (32.1756) | 0.0090 (22.8030) | 0.0032 (7.9026) | 0.0035 (28.6322) | 0.0032 (14.2298)

10. Secondary Outcome: Apparent Body Clearance (Cl/F)
Time Frame: as for outcome 2
Population: All randomized participants who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute CI/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour (L/h)
Arm/Group | 15 mg KQ-791 (Fasting) | 60 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fed) | 600 mg KQ-791 (Fasting) | 1200 mg KQ-791 (Fasting) | 1800 mg Kq-791 (Fasting)
Number analyzed (Participants) | 5 | 3 | 6 | 2 | 6 | 6 | 6
Liters per hour (L/h) | 0.3696 (48.4762) | 0.4666 (43.0267) | 0.5027 (32.8329) | 1.6219 (9.8091) | 0.7732 (47.0999) | 0.9150 (37.9245) | 0.8271 (40.4976)

11. Secondary Outcome: Apparent Volume of Distribution (Vd/F)
Time Frame: as for outcome 2
Population: All randomized participants who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute Vd/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | 15 mg KQ-791 (Fasting) | 60 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fed) | 600 mg KQ-791 (Fasting) | 1200 mg KQ-791 (Fasting) | 1800 mg Kq-791 (Fasting)
Number analyzed (Participants) | 5 | 3 | 6 | 2 | 6 | 6 | 6
Liters | 107.01 (34.95) | 132.23 (32.37) | 155.49 (27.72) | 179.83 (13.14) | 245.08 (46.56) | 261.06 (18.01) | 257.25 (29.61)

12. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-inf) in Fed Versus Fasting State
Time Frame: as for outcome 2
Population: All randomized participants who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute AUC0-inf in Fed versus Fasting State.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- 195 mg KQ-791: Food Effect (Fed/Fasting)
Arm/Group | 195 mg KQ-791
Number analyzed (Participants) | 2
h*ng/mL | 0.32 (15.17)

13. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Non-Zero Concentration (AUC0-t) in Fed Versus Fasting State
Time Frame: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 195 mg KQ-791
Number analyzed (Participants) | 6
h*ng/mL | 0.31 (37.61)

14. Secondary Outcome: Maximum Observed Drug Concentration (Cmax) in Fed Versus Fasting State
Time Frame: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 195 mg KQ-791
Number analyzed (Participants) | 6
ng/mL | 0.50 (59.94)

15. Secondary Outcome: Time to Maximum Drug Concentration (Tmax) in Fed Versus Fasting State
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8,10, 24, 48, 96, and 144 hours post-dose, and on Day 10 for all dose levels
Measure: Median (Full Range); unit: Hours
Arm/Group | 195 mg KQ-791
Number analyzed (Participants) | 6
Hours | 3 [-40.01 to 5.99]

16. Secondary Outcome: Amount of Drug Excreted in Urine
Time Frame: Four hour intervals up to 12 hours, and then 12-24 hours post dose
Population: All randomized participants who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute the Amount of Drug Excreted in Urine.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg
Groups:
- 15 mg KQ-791 (Fasting); 60 mg KQ-791 (Fasting); 195 mg KQ-791 (Fasting); 1200 mg KQ-791 (Fasting); 1800 mg Kq-791 (Fasting): 12-24 hours post-dose
- 195 mg KQ-791 (Fed); 600 mg KQ-791 (Fasting): 12-24 hours post dose
Arm/Group | 15 mg KQ-791 (Fasting) | 60 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fed) | 600 mg KQ-791 (Fasting) | 1200 mg KQ-791 (Fasting) | 1800 mg Kq-791 (Fasting)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 6
μg | 37.72 (27.71) | 155.51 (15.81) | 381.35 (34.71) | 224.51 (31.25) | 739.07 (67.68) | 1796.43 (29.85) | 3069.11 (37.08)

17. Secondary Outcome: Cumulative Urinary Excretion From Time Zero to Time t (Ae0-t)
Time Frame: Four hour intervals up to 12 hours, and then 12-24 hours post dose
Population: All randomized participants who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute Ae0-t.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg
Arm/Group | 15 mg KQ-791 (Fasting) | 60 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fed) | 600 mg KQ-791 (Fasting) | 1200 mg KQ-791 (Fasting) | 1800 mg Kq-791 (Fasting)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 6
μg | 90.60 (37.17) | 350.68 (19.39) | 859.41 (39.32) | 421.70 (27.23) | 1893.11 (57.89) | 3793.47 (34.98) | 6680.04 (38.34)

18. Secondary Outcome: Maximum Rate of Urinary Excretion (Rmax)
Time Frame: Four hour intervals up to 12 hours, and then 12-24 hours post dose
Population: All randomized participants who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute Rmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/hour
Arm/Group | 15 mg KQ-791 (Fasting) | 60 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fed) | 600 mg KQ-791 (Fasting) | 1200 mg KQ-791 (Fasting) | 1800 mg Kq-791 (Fasting)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
μg/hour | 5.13 (44.88) | 21.09 (29.33) | 49.05 (39.75) | 25.53 (29.88) | 123.11 (48.42) | 206.83 (33.25) | 377.72 (38.11)

19. Secondary Outcome: Time of Rmax Urinary Excretion (TRmax)
Time Frame: Four hour intervals up to 12 hours, and then 12-24 hours post dose
Population: All randomized participants who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute TRmax.
Measure: Median (Full Range); unit: Hours
Arm/Group | 15 mg KQ-791 (Fasting) | 60 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fed) | 600 mg KQ-791 (Fasting) | 1200 mg KQ-791 (Fasting) | 1800 mg Kq-791 (Fasting)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours | 5.93 [5.91 to 5.94] | 5.93 [5.90 to 9.91] | 5.91 [5.87 to 9.90] | 9.88 [5.85 to 9.91] | 5.88 [5.86 to 5.90] | 9.90 [5.84 to 9.96] | 5.96 [5.89 to 9.94]

20. Secondary Outcome: Renal Clearance (Clr)
Description: Calculated by the following equation: Ae0-t/AUC0-24
Time Frame: Four hour intervals up to 12 hours, and then 12-24 hours post dose
Population: All randomized participants who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute Clr.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | 15 mg KQ-791 (Fasting) | 60 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fed) | 600 mg KQ-791 (Fasting) | 1200 mg KQ-791 (Fasting) | 1800 mg Kq-791 (Fasting)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 6
Liters per hour | 0.0266 (31.5426) | 0.0286 (19.7181) | 0.0259 (19.7678) | 0.0252 (20.7044) | 0.0313 (17.2647) | 0.0333 (18.6140) | 0.0375 (9.5596)

ADVERSE EVENTS:
Description: Collected at each visit
Arm/Group | 15 mg KQ-791 (Fasting) | 60 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fasting) | 195 mg KQ-791 (Fed) | 600 mg KQ-791 (Fasting) | 1200 mg KQ-791 (Fasting) | 1800 mg Kq-791 (Fasting) | Placebo (Fasting) | Placebo (Fed)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/17 | 0/3
Other Adverse Events (participants affected / at risk) | 3/6 | 2/6 | 3/6 | 2/6 | 2/6 | 2/6 | 4/6 | 8/17 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 mg KQ-791 (Fasting) (N=6) | 60 mg KQ-791 (Fasting) (N=6) | 195 mg KQ-791 (Fasting) (N=6) | 195 mg KQ-791 (Fed) (N=6) | 600 mg KQ-791 (Fasting) (N=6) | 1200 mg KQ-791 (Fasting) (N=6) | 1800 mg Kq-791 (Fasting) (N=6) | Placebo (Fasting) (N=17) | Placebo (Fed) (N=3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Faeces discolored (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastresophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood tryglycerides increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Blood pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
High density lipoprotein decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart Rate Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Protein urine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increases (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other